CLINICAL TRIAL: NCT03279965
Title: A Pilot Study to Assess the Use of MRI in the Assessment of Patients With Cystic Fibrosis and Primary Ciliary Dyskinesia
Brief Title: MRI in Cystic Fibrosis and Primary Ciliary Dyskinesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Bioxydyn Ltd, Manchester (Unknown); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016LI002B
Record Dates: First submitted 2017-06-19; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis; Primary Ciliary Dyskinesia
Keywords: Lung MRI cystic fibrosis primary ciliary dyskinesia
MeSH Terms: conditions — Cystic Fibrosis; Ciliary Motility Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis: Patients with known cystic fibrosis
  Interventions: Diagnostic Test: MRI
- Primary ciliary dyskinesia: Patients with known primary ciliary dyskinesia
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI of lungs, paranasal sinuses and liver in addition to established clinical examinations (lung CT, pulmonary function testing)
  Other Names: Nuclear magnetic resonance (NMR)

SUMMARY:
This is a small pilot / feasibility study (Approximately 50 patients) to assess the possibility of clinical implementation of MRI assessment of patients with cystic fibrosis and primary ciliary dyskinesia.

Patients will undergo their standard CT imaging and lung function investigations and additionally will undergo MRI examination. Reports from CT (the current gold standard) and MRI will be assessed for concordance and patient acceptability and examination implementation costs will also be assessed. Novel MRI-based potential markers of CF and PCD disease state will also be assessed.

DETAILED DESCRIPTION:
In this small single site pilot / feasibility study we aim to recruit approximately 50 patients over the age of 6 years with known cystic fibrosis (CF) or primary ciliary dyskinesia (PCD).

Patients will be recruited from routine clinic appointments or at admission for inpatient investigation and/or treatment at the point of referral for computed tomography (CT) examination. If they consent to participation they will undergo MRI examination in addition to their standard clinical CT (within 7 days of the CT scan - on the same day if practicable).

The magnetic resonance imaging (MRI) scans will be anonymised and reported by radiologists, blinded to the CT findings. The reports and scores (Eichinger and Brody2) will then be compared those of the standard CT to assess concordance between the modalities and inter and intra observer variability.

Potential novel biomarkers (pulmonary ventilation and perfusion (non-contrast) and sinus mucus and liver tissue characteristics) will be compared with established markers (including lung clearance index) and known CF mutation / PCD type.

Patients or their carers will also be asked to fill in a short questionnaire comparing the differential patient acceptability of CT and MRI examinations. The cost (time, resources etc) of each examination will be calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Known CF or PCD Referred for CT chest

Exclusion Criteria:

* Contraindication to MRI (Pacemaker etc) Unable to stay still for MRI

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known cystic fibrosis or primary ciliary dyskinesia referred for CT chest as part of routine outpatient or inpatient investigations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-05-05 (Estimated); Study Completion 2018-05-05 (Estimated)

PRIMARY OUTCOMES:
Structural and quantitative MRI vs CT in cystic fibrosis and primary ciliary dyskinesia assessment | 18 months
  To determine whether MRI with ventilation imaging can produce sufficiently diagnostic images, in the setting of CF or PCD, to replace CT imaging follow up. This will be assessed via semi-quantitative visual scoring (CT-based Brody / CFCT score and MRI-based Eichinger score) with both scoring systems applied to both CT and MRI. Scoring of the "air-trapping" component of CFCT will be substituted with scoring of ventilation defects on MRI. Scores will come from 2 observers, blinded to each others opinion, with a 3rd observer acting to resolve discrepancies. Intermodality variation will be assessed via ICC and Bland-Altman

SECONDARY OUTCOMES:
Ventilation MRI vs Lung clearance index (LCI) | 18 months
  Dynamic oxygen enhanced MRI measures will be compared to equivalent measurements from lung clearance testing. Bland Altman and ICC analysis of time to oxygen wash in (in seconds) on MRI, to time to nitrogen washout in seconds from lung clearance testing
Sinus disease and exacerbations 1 | 18 months
  Simple correlative statistics of degree of sinus opacification (percentage volume occupied by mucus and polyps) with frequency of infective exacerbations (number per month)
Sinus disease and exacerbations 2 | 18 months
  Simple correlative statistics of degree of sinus opacification (percentage volume occupied by mucus and polyps) with rate of decline in spirometry measures (percentage drop in predicted FEV1 and FEV1/FVC over the 6 months prior to scanning)
Sinus disease and exacerbations 3 | 18 months
  Simple correlative statistics of presence of susceptibility artefact in sinus mucus (binary; yes, no) with micro-organism cultured (nominal)
Liver disease 1 | 18 months
  Simple correlation of liver volume (cm3) and T1 relaxation time (ms) with serologic markers of liver function (AST, ALT and ALP in IU/L and albumin in g/L)
Liver disease 2 | 18 months
  Simple correlation of liver T1 relaxation time (ms) with ultrasound elastography markers of liver fibrosis (sheer wave speed in m/s)
Patient acceptability | 18 months
  To determine whether MRI is as acceptable to patients with CF or PCD as CT. This is via simple descriptive statistics from a bespoke questionnaire consisting of 5-point Likert scale questions regarding each scan.
Clinical implementation | 18 months
  To determine the operational cost differences in implementing MRI follow up vs CT follow up. Simple comparison of cost (in GBP) of diagnostic CT vs lung MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Devaraj, Principal Investigator — Royal Brompton Hospital, London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data outside the research team at this time.